CLINICAL TRIAL: NCT02954185
Title: Wellclub Shoulder Therapy Outcome Validation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment/Financial Issues
Sponsor: University of Minnesota (Other)
Collaborators: Fairview Sports Physical Therapy Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1607M91681
Record Dates: First submitted 2016-10-07; First posted 2016-11-03 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Shoulder Pain
Keywords: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WellClub Device (Experimental): Hand held device that patients use for home therapy
  Interventions: Other: WellClub
- Standard Therapy (Active Comparator): Standard care therapy for should pain
  Interventions: Behavioral: Standard Therapy

INTERVENTIONS:
Other: WellClub
  Arms: WellClub Device
Behavioral: Standard Therapy
  Arms: Standard Therapy

SUMMARY:
Preliminary evaluations have been completed and resulted in patients and therapist indicating positive outcomes through increased patient engagement, asynchronous communications (i.e. messaging) between therapists and patients, and objective assessment and monitoring of exercises performed by the patients. The investigator's hypothesis is that patients using the Wellclub device and application in addition to in-clinic physical therapy will be more compliant with their home exercise programs and have the same or better functional outcomes than patients with similar conditions who use in-clinic care only.

DETAILED DESCRIPTION:
Patients seeking an initial outpatient physical therapy evaluation for non-surgical shoulder impingement with pain, who own iPhones with iOS 8 or later. Patients will be randomized into the study group or the control group, and be seen at least once per week by their physical therapist for the duration of the therapy episode, or up to 12 weeks. The study group will be asked to strap to their wrist a small, measurement device and download a smartphone application. The App communicates with the wearable device and reminds them to complete their therapy and provides patients visual instruction, feedback on exercise quality, and exercise count for the prescribed physical therapy. The control group will only have traditional in-clinic therapy as deemed clinically necessary by the PT.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder impingement not requiring immediate surgery

Exclusion Criteria:

* Rotator cuff tear (RCT)
* Surgical history of rotator cuff repair (RCR)
* Cortisone injection or other injectable for past 6 months
* Prescription NSAIDs in the past 6 months
* Frozen shoulder syndrome
* Neurological conditions
* Other orthopaedic conditions (spine/neck)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Change in performance measured by percentages | Baseline and 6 weeks
  Percentage of completed exercises correctly completed by the patient
Change in score on SPADI (Shoulder Pain And Disability Index) | Baseline and 6 weeks
  SPADI is a scale consisting of 0-10 0 being the best and 10 being the worse pain ever
Change in degrees of shoulder range of motion | Baseline and 6 weeks
  Change in range of motion on metered scale

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ames, PT PhD, Principal Investigator — Fairview Sports Physical Therapy Program
Locations (5):
- United States (5):
  - Fairview - Institute for Athletic Medicine, Blaine, Minnesota
  - Fairview - Institute for Athletic Medicine, Eden Prairie, Minnesota
  - Fairview - Institute for Athletic Medicine, Edina, Minnesota
  - University Orthopaedic Therapy Center, Minneapolis, Minnesota
  - Fairview - Institute for Athletic Medicine, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided